CLINICAL TRIAL: NCT00858208
Title: Long-Term Non-Interventional Study To Investigate The Efficacy And Safety Of MACUGEN In Patients With Neovascular Age-Related Macular Degeneration Under Conditions Of Routine Clinical Practice.
Brief Title: Efficacy And Safety Of Macugen In Patients With Neovascular AMD In Routine Clinical Practice.
Acronym: MACULA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5751028
Record Dates: First submitted 2009-02-26; First posted 2009-03-09 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2011-09

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: efficacy and safety of Macugen in routine clinical practice
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with neovascular Age-Related Macula Degeneration
  Interventions: Drug: pegaptanib sodium

INTERVENTIONS:
Drug: pegaptanib sodium — pegaptanib sodium intravitreal injection every 6 weeks for 2 years

SUMMARY:
Efficacy and safety of MACUGEN in patients suffering from neovascular age-related macular degeneration in routine clinical practice at least as good as demonstrated in randomized multicenter clinical trials.

DETAILED DESCRIPTION:
Eligible patients in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

adults with neovascular age-related macula degeneration

Exclusion Criteria:

according to SmPC

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Age-related Macula degeneration
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Greece (7):
  - Pfizer Investigational Site, Pátrai, Pellopoese
  - Pfizer Investigational Site, Alexandroupoli
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Larissa
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
  - Pfizer Investigational Site, Xánthi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751028&StudyName=Efficacy%20And%20Safety%20Of%20Macugen%20In%20Patients%20With%20Neovascular%20AMD%20In%20Routine%20Clinical%20Practice.

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegaptanib: The usage and dosage recommendations for Macugen (Pegaptanib) was in accordance with the local Summary of Product Characteristics. Participants received Pegaptanib in one eye (designated study eye) while the fellow eye did not receive Pegaptanib.
Period: Overall Study
Arm/Group | Pegaptanib
Started | 85
Completed | 6
Not Completed | 79
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 26
Not completed — Participant refused | 40
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Arm/Group | Pegaptanib
Number analyzed (Participants) | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 74.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 41
National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) sub-scale scores at baseline [Mean (Standard Deviation); unit: scores on a scale] — Participant-reported 25 item questionnaire. Responses to each question converted to 0-100 score. Questions grouped into 11 vision-targeted categories and 1 general heath category. Sub-scale score=mean score in a category. Range of sub-scale scores=0 to 100 where higher scores represent better functioning. n=participants with evaluable data.
  scores on a scale
    General Health (n=85) | 45.00 (23.081)
    General Vision (n=85) | 55.53 (16.439)
    Ocular Pain (n=85) | 80.74 (20.912)
    Near Activities (n=85) | 53.09 (28.976)
    Distance Activities (n=85) | 58.73 (28.264)
    Social Functioning (n=85) | 72.35 (28.809)
    Mental Health (n=85) | 50.51 (24.056)
    Role Difficulties (n=85) | 57.06 (31.425)
    Dependency (n=85) | 61.27 (28.542)
    Driving (n=30) | 49.72 (35.523)
    Color Vision (n=83) | 79.82 (23.896)
    Peripheral Vision (n=85) | 67.65 (29.586)
Procedures used for age-related macular degeneration (AMD) diagnosis [Number; unit: participants] — Procedures used in the diagnosis of age-related macular degeneration (AMD) included fluorescein angiography, indocyanine green angiography, and optical coherence tomography.
  participants
    fluorescein angiography | 66
    indocyanine green angiography | 0
    optical coherence tomography | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Visual Acuity (VA) at the Final Visit
Description: VA measured using Early Treatment Diabetic Retinopathy Study (ETDRS), Snellen chart, or other methods verifying if the participant was able to count fingers, perceive hand motion, or light. VA expressed as the logarithm of the minimum angle of resolution (logMAR), and could range from 0 (representing 20/20 vision) to 1. Change: VA Score at Visit X minus VA Score at Baseline, where a negative change in the logMAR scale represents an improvement in VA.
Time Frame: Baseline, Week 102 or Early Termination (ET)
Population: Safety Analysis Set (SAS) = Full Analysis Set (FAS): Enrolled participants who received at least 1 dose of Pegaptanib; Number of participants analyzed (N)=participants with evaluable data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 67
Number analyzed (eyes) | 67
logMAR
  Baseline | 0.829 (0.367)
  Change at Week 102/ET | -0.126 (0.371)
Statistical Analysis 1: Comparison: Pegaptanib; Test type: Superiority or Other; p = 0.0072, paired t-test

2. Secondary Outcome: Change From Baseline VA at Each Visit
Description: as for outcome 1
Time Frame: Baseline, every 6 weeks up to Week 102
Population: SAS; Number of participants analyzed (N)=participants with evaluable data; n=participants with evaluable data at specified time point
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 67
Number analyzed (eyes) | 67
logMAR
  Change at Week 6 (n=59) | -0.07 (0.249)
  Change at Week 12 (n=56) | -0.10 (0.297)
  Change at Week 18 (n=48) | -0.12 (0.374)
  Change at Week 24 (n=43) | -0.16 (0.406)
  Change at Week 30 (n=37) | -0.16 (0.415)
  Change at Week 36 (n=31) | -0.17 (0.416)
  Change at Week 42 (n=28) | -0.12 (0.455)
  Change at Week 48 (n=25) | -0.13 (0.472)
  Change at Week 54 (n=23) | -0.07 (0.461)
  Change at Week 60 (n=19) | -0.09 (0.500)
  Change at Week 66 (n=13) | 0.04 (0.558)
  Change at Week 72 (n=10) | 0.05 (0.495)
  Change at Week 84 (n=8) | -0.04 (0.302)
  Change at Week 90 (n=4) | -0.11 (0.334)
  Change at Week 96 (n=2) | 0.33 (0.213)
  Change at Week 102 (n=2) | 0.33 (0.213)
Statistical Analysis 1: Comparison: Pegaptanib; Change from baseline at Week 6; Test type: Superiority or Other; p = 0.0433, paired t-test
Statistical Analysis 2: Comparison: Pegaptanib; Change from baseline at Week 12; Test type: Superiority or Other; p = 0.0133, paired t-test
Statistical Analysis 3: Comparison: Pegaptanib; Change from baseline at Week 18; Test type: Superiority or Other; p = 0.0278, paired t-test
Statistical Analysis 4: Comparison: Pegaptanib; Change from baseline at Week 24; Test type: Superiority or Other; p = 0.0160, paired t-test
Statistical Analysis 5: Comparison: Pegaptanib; Change from baseline at Week 30; Test type: Superiority or Other; p = 0.0264, paired t-test
Statistical Analysis 6: Comparison: Pegaptanib; Change from baseline at Week 36; Test type: Superiority or Other; p = 0.0278, paired t-test
Statistical Analysis 7: Comparison: Pegaptanib; Change from baseline at Week 42; Test type: Superiority or Other; p = 0.1854, paired t-test
Statistical Analysis 8: Comparison: Pegaptanib; Change from baseline at Week 48; Test type: Superiority or Other; p = 0.1684, paired t-test
Statistical Analysis 9: Comparison: Pegaptanib; Change from baseline at Week 54; Test type: Superiority or Other; p = 0.4718, paired t-test
Statistical Analysis 10: Comparison: Pegaptanib; Change from baseline at Week 60; Test type: Superiority or Other; p = 0.4340, paired t-test
Statistical Analysis 11: Comparison: Pegaptanib; Change from baseline at Week 66; Test type: Superiority or Other; p = 0.7765, paired t-test
Statistical Analysis 12: Comparison: Pegaptanib; Change from baseline at Week 72; Test type: Superiority or Other; p = 0.7544, paired t-test
Statistical Analysis 13: Comparison: Pegaptanib; Change from baseline at Week 84; Test type: Superiority or Other; p = 0.7201, paired t-test
Statistical Analysis 14: Comparison: Pegaptanib; Change from baseline at Week 90; Test type: Superiority or Other; p = 0.5692, paired t-test
Statistical Analysis 15: Comparison: Pegaptanib; Change from baseline at Week 96; Test type: Superiority or Other; p = 0.2749, paired t-test
Statistical Analysis 16: Comparison: Pegaptanib; Change from baseline at Week 102; Test type: Superiority or Other; p = 0.2749, paired t-test

3. Secondary Outcome: Change From Baseline VA at the Final Visit for Participants With Vascular Retinal Pigment Epithelial Detachment (RPED)
Description: VA measured using Early Treatment Diabetic Retinopathy Study (ETDRS), Snellen chart, or other methods verifying if the participant was able to count fingers, perceive hand motion, or light. VA expressed as the logarithm of the minimum angle of resolution (logMAR), and could range from 0 (representing 20/20 vision) to 1. Change: VA Score at Visit X minus VA Score at Baseline, where a negative change in the logMAR scale represents an improvement in VA. On the case report form, participants with RPED=those with the "Pigment Epithelial Detachment (PED) present" box ticked at Baseline Visit.
Time Frame: Baseline, Week 102 or ET
Population: SAS subset of participants with RPED at baseline
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 28
Number analyzed (eyes) | 28
logMAR
  Baseline | 0.804 (0.386)
  Change at Week 102/ET | -0.105 (0.443)

4. Secondary Outcome: Change From Baseline NEI-VFQ-25 Overall Composite Score at Each Visit
Description: Participant-reported 25 item questionnaire. Responses to each question converted to 0-100 score. Questions grouped into 11 vision-targeted categories and 1 general health category. Mean score calculated for each category. Overall composite score=mean of 11 vision-targeted sub categories. Range of composite score=0 to 100 where higher scores represent better functioning. Change: Composite score at Visit X minus composite Score at Baseline, where higher scores represent better functioning.
Time Frame: Baseline, Month 6, 12, 18, and 24
Population: SAS; N=participants with evaluable data; n=participants with evaluable data at specified time point
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pegaptanib
Number analyzed (Participants) | 30
scores on a scale
  Baseline (n=30) | 67.73 (21.126)
  Change at Month 6 (n=19) | 2.62 (10.647)
  Change at Month 12 (n=13) | 4.22 (9.596)
  Change at Month 18 (n=4) | -2.33 (1.549)
  Change at Month 24 (n=2) | -2.56 (9.241)
Statistical Analysis 1: Comparison: Pegaptanib; Change at Month 6; Test type: Superiority or Other; p = 0.2970, paired t-test
Statistical Analysis 2: Comparison: Pegaptanib; Change at Month 12; Test type: Superiority or Other; p = 0.1392, paired t-test
Statistical Analysis 3: Comparison: Pegaptanib; Change at Month 18; Test type: Superiority or Other; p = 0.0573, paired t-test
Statistical Analysis 4: Comparison: Pegaptanib; Change at Month 24; Test type: Superiority or Other; p = 0.7625, paired t-test

5. Secondary Outcome: Change From Baseline NEI-VFQ-25 Overall Composite Score at Final Visit
Description: as for outcome 4
Time Frame: Baseline, Week 102 or ET
Population: SAS; N=participants with evaluable data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pegaptanib
Number analyzed (Participants) | 20
scores on a scale
  Baseline | 69.47 (21.62)
  Change at Week 102/ET | 3.21 (12.78)
Statistical Analysis 1: Comparison: Pegaptanib; Test type: Superiority or Other; p = 0.2759, paired t-test

6. Secondary Outcome: Change From Baseline NEI-VFQ-25 Sub-scale Scores at Final Visit
Description: Participant-reported 25 item questionnaire. Responses to each question converted to 0-100 score. Questions grouped into 11 vision-targeted categories and 1 general heath category. Sub-scale score=mean score in a category. Range of sub-scale scores=0 to 100 where higher scores represent better functioning. Change: Sub-scale scores score at Visit X minus sub-scale score at Baseline, where higher scores represent better functioning.
Time Frame: Baseline, Week 102 or ET
Population: SAS; N=participants with evaluable data; n=participants with evaluable data at specified time point and item in questionnaire
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pegaptanib
Number analyzed (Participants) | 85
scores on a scale
  General Health, Change at Week 102/ET (n=59) | -1.69 (22.198)
  General Vision, Change at Week 102/ET (n=59) | 5.08 (16.014)
  Ocular Pain, Change at Week 102/ET (n=59) | -4.87 (15.746)
  Near Activities, Change at Week 102/ET (n=59) | 5.93 (21.709)
  Distance Activities, Change at Week 102/ET (n=59) | 0.71 (20.532)
  Social Functioning, Change at Week 102/ET (n=59) | 1.91 (22.602)
  Mental Health, Change at Week 102/ET (n=59) | 3.81 (18.461)
  Role Difficulties, Change at Week 102/ET (n=59) | 4.45 (17.794)
  Dependency, Change at Week 102/ET (n=59) | 6.07 (18.751)
  Driving, Change at Week 102/ET (n=20) | -2.50 (14.075)
  Color Vision, Change at Week 102/ET (n=57) | 3.07 (20.084)
  Peripheral Vision, Change at Week 102/ET (n=59) | 5.08 (19.575)

7. Other Pre Specified Outcome: Change From Baseline VA at Final Visit by Age Group
Description: Participant population (by age group) that benefited more from Pegaptanib treatment based on change from baseline VA at final visit. VA measured by age group (51 to 64 years, greater than or equal to [>=] 65 years) using ETDRS chart at 4 meter distance, at 1 meter distance (if participant's VA was poor) or verifying if participant able only to count fingers, perceive hand motion, or light. VA expressed as logMAR could range from 0 (representing 20/20 vision) to 1. Change: VA Score at Visit X minus VA Score at Baseline, where a negative change in logMAR scale represents improvement in VA.
Time Frame: Baseline, Week 102 or ET
Population: SAS;N=participants with evaluable data; n=participants with evaluable data at specified time point and age group
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 67
Number analyzed (eyes) | 67
logMAR
  51-64 years, Baseline (n=10) | 0.797 (0.361)
  51-64 years, Change at Week 102/ET (n=10) | -0.156 (0.253)
  ≥ 65 years, Baseline (n=57) | 0.835 (0.371)
  ≥ 65 years, Change at Week 102/ET (n=57) | -0.121 (0.390)

8. Other Pre Specified Outcome: Change From Baseline VA at the Final Visit by Age-related Macular Degeneration (AMD) Stage
Description: Participant population (by AMD stage) that benefited more from Pegaptanib treatment based on change from baseline VA at final visit. VA measured by AMD stage (early lesion, late stage lesion, other) using ETDRS chart at 4 meter distance, at 1 meter distance (if participant's VA was poor) or verifying if participant able only to count fingers, perceive hand motion, or light. VA expressed as logMAR could range from 0 (representing 20/20 vision) to 1. Change: VA Score at Visit X minus VA Score at Baseline, where a negative change in logMAR scale represents improvement in VA.
Time Frame: Baseline, Week 102 or ET
Population: SAS subset of participants with AMD; n=participants with evaluable data at specified time point and stage of AMD
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 66
Number analyzed (eyes) | 66
logMAR
  Early Lesion, Baseline (n=34) | 0.704 (0.332)
  Early Lesion, Change at Week 102/ET (n=34) | -0.066 (0.395)
  Late Stage Lesion, Baseline (n=31) | 0.961 (0.358)
  Late Stage Lesion, Change at Week 102/ET (n=31) | -0.190 (0.348)
  Other AMD Stage, Baseline (n=1) | 1.301 (NA) — Not Available (NA): only 1 participant with data
  Other AMD Stage, Change at Week 102/ET (n=1) | -0.301 (NA) — Only 1 participant with data

9. Other Pre Specified Outcome: Change From Baseline VA at the Final Visit by Previous Treatment of AMD
Description: Participant population (by previous treatment of AMD) that benefited more from Pegaptanib treatment based on change from baseline VA at final visit. VA measured by previous AMD treatment (yes/no) using ETDRS chart at 4 meter distance, at 1 meter distance (if participant's VA was poor) or verifying if participant able only to count fingers, perceive hand motion, or light. VA expressed as logMAR could range from 0 (representing 20/20 vision) to 1. Change: VA Score at Visit X minus VA Score at Baseline, where a negative change in logMAR scale represents improvement in VA.
Time Frame: Baseline, Week 102 or ET
Population: SAS subset of participants for who data was collected about previous AMD treatment (yes/no); n=number of participants with evaluable data at specified time point
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 67
Number analyzed (eyes) | 67
scores on a scale
  No Previous AMD Treatment, Baseline (n=62) | 0.838 (0.363)
  No Previous Treatment, Change at Week 102/ET(n=62) | -0.126 (0.367)
  Previous AMD Treatment, Baseline (n=5) | 0.724 (0.438)
  Previous Treatment, Change at Week 102/ET (n=5) | -0.120 (0.461)

10. Other Pre Specified Outcome: Number of Participants for Whom Fluorescein Angiography Was Used to Monitor the Course of AMD Treatment
Description: Participant counts by type of diagnostic procedure (fluorescein angiography) used to monitor AMD treatment.
Time Frame: Every 6 weeks up to Week 102
Population: SAS
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 85
participants
  Week 6 | 8
  Week 12 | 7
  Week 18 | 6
  Week 24 | 7
  Week 30 | 11
  Week 36 | 4
  Week 42 | 3
  Week 48 | 4
  Week 54 | 2
  Week 60 | 4
  Week 66 | 2
  Week 72 | 0
  Week 78 | 0
  Week 84 | 1
  Week 90 | 1
  Week 96 | 0
  Week 102 | 1

11. Other Pre Specified Outcome: Number of Participants for Whom Optical Coherence Tomography Was Used to Monitor the Course of AMD Treatment
Description: Participant counts by type of diagnostic procedure (optical coherence tomography) used to monitor AMD treatment.
Time Frame: Every 6 weeks up to Week 102
Population: SAS
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 85
participants
  Week 6 | 32
  Week 12 | 35
  Week 18 | 34
  Week 24 | 31
  Week 30 | 24
  Week 36 | 26
  Week 42 | 21
  Week 48 | 17
  Week 54 | 16
  Week 60 | 16
  Week 66 | 10
  Week 72 | 6
  Week 78 | 0
  Week 84 | 7
  Week 90 | 5
  Week 96 | 1
  Week 102 | 1

12. Other Pre Specified Outcome: Number of Participants for Whom Indocyanine Green Angiography Was Used to Monitor the Course of AMD Treatment
Description: Participant counts by type of diagnostic procedure (indocyanine green angiography) used to monitor AMD treatment.
Time Frame: Every 6 weeks up to Week 102
Population: SAS
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 85
participants
  Week 6 | 0
  Week 12 | 0
  Week 18 | 0
  Week 24 | 0
  Week 30 | 0
  Week 36 | 1
  Week 42 | 0
  Week 48 | 0
  Week 54 | 0
  Week 60 | 0
  Week 66 | 0
  Week 72 | 0
  Week 78 | 0
  Week 84 | 0
  Week 90 | 0
  Week 96 | 0
  Week 102 | 0

13. Other Pre Specified Outcome: Number of Participants Who Discontinued Treatment Prematurely or Changed Treatment During the Course of the Study
Description: Participants with dose reduction or temporary discontinuation of treatment due to adverse events (AEs).
Time Frame: Baseline through Week 102
Population: SAS
Measure: Number; unit: participants
Arm/Group | Pegaptanib
Number analyzed (Participants) | 85
participants | 3

14. Other Pre Specified Outcome: Change From Baseline to Final Visit in Intraocular Pressure (IOP) (Before and After Injection)
Description: IOP was measured using either applanation or tonopen before intravitreal injection, reported as pre-dose and post-dose pressure. IOP valid range: 10-21 mmHg. Change: IOP at Visit X minus IOP at Baseline.
Time Frame: Baseline and Week 102 or ET
Population: SAS; N=participants with evaluable data at baseline; n=participants with evaluable data at specified time point
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Units Other Than Participants: eyes
Arm/Group | Pegaptanib
Number analyzed (Participants) | 78
Number analyzed (eyes) | 78
millimeters of mercury (mmHg)
  Baseline (n=78) | 15.0 (3.2)
  Pre-dose, Change at Week 102/ET (n=74) | 0.3 (2.7)
  Post-dose, Change at Week 102/ET (n=75) | 0.8 (3.1)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pegaptanib
Serious Adverse Events (participants affected / at risk) | 1/85
Other Adverse Events (participants affected / at risk) | 5/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegaptanib (N=85)
Intestinal polyp (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegaptanib (N=85)
Retinal tear (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Asthenia (General disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.